CLINICAL TRIAL: NCT00949169
Title: Association of Carotid IMT and Large-vessel Atherosclerosis by MDCT in Korean Type 2 Diabetic Patients
Brief Title: Carotid Intima-media Thickness (IMT) and Large-vessel Atherosclerosis by Multidetector Computed Tomography (MDCT)
Status: Completed | Type: Observational
Sponsor: Eulji University Hospital (Other)
Responsible Party: Department of Internal Medicine, Eulji University Hospital
Other Study IDs: Eulji07-34
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Type 2 Diabetes
Keywords: Atherosclerosis; Carotid IMT; Multidetector CT; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Carrotid IMT group according to maximal IMT: We defined increased IMT group as whom had maximal IMT ≥ 1.0 mm.

SUMMARY:
The aim of this study was to investigate whether carotid IMT can predict the presence of more advanced atherosclerosis such as carotid stenosis, coronary or intracranial artery disease by MDCT and whether MDCT could be useful next step for more aggressive treatment modality in Korean type 2 diabetic patients.

DETAILED DESCRIPTION:
We evaluated mean/maximal carotid IMT in seventy-one type 2 diabetic subjects, and defined increased carotid IMT as maximal IMT ≥ 1.0 mm. Multidetector CT (MDCT) and pulse wave velocity (PWV) were taken to evaluate carotid artery stenosis (CS), coronary artery disease (CAD), intracranial arterial lesion (ICA), and peripheral artery disease (PAD). We compared prevalence of large artery stenosis according to carotid IMT group and evaluated whether maximal IMT ≥ 1.0 mm could predict for significant CAD by MDCT. We performed invasive coronary angiography in some patients (N=14) and analyzed association for degrees of CAD between two angiographic methods.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients who had multiple cardiovascular risk factors were recruited.
* Patients who had atypical chest pain, EKG abnormality (ischemic ST-T changes or abnormal Q-wave), or history of previous cardiovascular disease were also included.

Exclusion Criteria:

* Acute coronary SD, serum Cr>1.4 mg/dL, history of allergy to iodinated contrast dye were excluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetic patients who had multiple cardiovascular risk factors
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2006-04; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
We compared prevalence of large artery stenosis according to carotid IMT group and evaluated whether maximal IMT ≥ 1.0 mm could predict for significant CAD by MDCT. | 17 months

SECONDARY OUTCOMES:
We performed invasive coronary angiography in some patients (N=14) and analyzed association for degrees of CAD between two angiographic methods. | 17 months

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Wan Min, MD., PhD., Principal Investigator — Department of Internal Medicine, Eulji University Hospital
Locations (1):
- Eulji University Hospital, Seoul, South Korea